CLINICAL TRIAL: NCT00377494
Title: A Phase I Trial of PFCSP DNA/MVA.CSO Prime/Boost Vaccine in Mampong, Ghana
Brief Title: CS DNA MVA Trial in Mampong, Ghana
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-070; NMIMR: CPN 042/03-04
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2007-02

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: malaria, Plasmodium falciparum, vaccine, Ghana
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Vaccines

INTERVENTIONS:
Biological: MVA-CSO Vaccine
Biological: PfCSP DNA (VCL-2510) Vaccine

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and effectiveness of 2 doses of a malaria vaccine (DNA) followed by a dose of another type of malaria vaccine (MVA) given as a "booster." Forty-eight adults in Ghana, ages 18-50 years, will participate for 17 months. They will be randomly assigned to 1 of 4 treatment groups. Group 1 will receive the DNA malaria vaccine at months 0 and 1, and the booster at month 7. Group 2 will receive a rabies vaccine at months 0 and 1, and an injection containing no vaccine at month 7. Group 3 will receive the DNA malaria vaccine at months 5 and 6, and the booster at month 7. Group 4 will receive the rabies vaccine at months 5 and 6, and an injection containing no vaccine at month 7. Blood samples and information regarding health problems that may occur after vaccination will be collected.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, tolerability, and immunogenicity of immunization with 2 doses of the PfCSP DNA vaccine (given 1 month apart) followed by a single dose of MVA.CSO (given either 1 month or 6 months later) when administered to healthy, malaria semi-immune adult volunteers. This Phase 1, randomized study conducted at Tetteh Quarshie Memorial Hospital will enroll 48 healthy volunteers, ages 18 to 50 years. Twenty four volunteers will initially be recruited and randomized to Groups 1 and 2. During Months 4 and 5 of the study, another 24 volunteers will be recruited and randomized to Groups 3 and 4. Group 1 will receive the DNA malaria vaccine intramuscularly (IM) at months 0 and 1, and the MVA malaria vaccine intradermally (ID) at month 7. Group 2 will receive a rabies vaccine IM at months 0 and 1, and a normal saline injection ID at month 7. Group 3 will receive the DNA malaria vaccine IM at months 5 and 6, and the MVA malaria vaccine ID at month 7. Group 4 will receive the rabies vaccine IM at months 5 and 6, and a normal saline injection ID at month 7. Blood samples will be collected at intervals for safety and immunogenicity studies. Vaccine safety will be monitored until 10 months after the final dose. At the conclusion of the study, volunteers randomized to Groups 1 and 3 will have the option of receiving the rabies vaccine. The primary study objectives are to: (1) assess the safety and tolerability of immunization with two doses of PfCSP DNA followed by one dose of MVA.CSO in healthy, malaria semi-immune adult volunteers when given at intervals of 0, 1, and 2 months or at 0, 1, and 7 months; (2) evaluate whether the PfCSP DNA/MVA.CSO prime/boost vaccine regimen induces PfCSP-specific immune responses, as assessed by IFN-gamma ELISPOT assay, over background responses; and (3) evaluate whether extending the interval between the second dose of PfCSP DNA and MVA.CSO from 1 month to 6 months is associated with higher levels of PfCSP specific T cell responses in semi-immune adults. The secondary study objective is to evaluate whether extending the interval between the second dose of PfCSP DNA and MVA.CSO from 1 month to 6 months is associated with higher levels of humoral immunity by ELISA and IFAT in semi-immune adults. The principal outcome measure will be the incidence of any vaccine related adverse event, abnormal lab values, and local or systemic reactions. An additional outcome variable for the remaining primary objectives is the results of the IFN-gamma ELISPOT assay at 1 week after administration of MVA.CSO. This study is planned to be the first of multiple clinical trials designed to test malaria vaccines in adults, children, and infants in endemic regions of Ghana.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults, 18-50 years of age.
2. Available to participate for the duration of the study period.
3. HIV seronegative, per written proof of assay collected within four weeks of screening
4. Provision of personal (not proxy) agreement to consent to the study.

Exclusion Criteria:

1. Females who are pregnant or nursing, who plan on becoming pregnant or plan to nurse during the study period, or males who plan on fathering children during the study period.
2. Have a history of diabetes or any cardiovascular disorder
3. Have hypertension, or current treatment with anti-hypertensives.
4. Have a total cholesterol >197.5 mg/dL.
5. Have an abnormal EKG (e.g., all kinds of atrioventricular or intraventricular conditions or blocks such as complete left or right bundle branch block, A-V node block, QTc or PR prolongation, premature atrial contractions or other atrial arrhythmia, sustained ventricular arrhythmia, or 2 premature ventricular contractions (PVC) in a row, or ST elevation consistent with ischemia).
6. Have an abnormal Troponin I level.
7. Are HIV positive or have any known immunodeficiency (including receiving immunosuppressive therapy or a history of splenectomy).
8. Have a history of autoimmune disease (including inflammatory bowel disease, hemolytic anemia, autoimmune hepatitis, rheumatoid arthritis, lupus, etc.)
9. Have or have had any other illness or condition which, in the investigator's judgment, will substantially increase the risk associated with their participation or will compromise the scientific objectives of the protocol.
10. Have eczema/atopic dermatitis or other significant skin condition.
11. Have anemia, defined by a hemoglobin level < 12.7g/dl in males, and < 10.5 g/dl in females.
12. Have a creatinine level >141.2 mmol/L (males) or >120.5 mmol/L (females).
13. Have an ALT value >53.1 U/L in males, or >39.2 U/L in females.
14. Have an AST value >65.0 U/L in males, or >46.5 U/L in females.
15. Have a total bilirubin value > 1.4 mg/L
16. Have an alkaline phosphatase level > 297.8 U/L in males, or > 255.4 U/L in females.
17. Have a white cell count <3.4 x 10(9th)/L or > 8.8 x 10(9th)/L.
18. Have a platelet count <97.0 x 10(9th)/L in males, or <118.0 x 10(9th)/L in females
19. Have the presence of any glucose or greater than trace amounts of protein in the urine. Have the presence of greater than trace amounts of RBC in the urine of males and non-menstruating females.
20. Plan to have surgery between enrollment and the last immunization.
21. Have any known allergic reactions or hypersensitivity to any vaccinations in the past.
22. Decision to participate in another investigational vaccine/drug research during the period of this study.
23. Have any immunizations planned within three weeks of one of the study immunizations.
24. Receipt of immunoglobulins or any blood products within three months preceding the initial study immunization or planned administration during the study period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2008-07

CONTACTS AND LOCATIONS:
Locations (2):
- Naval Medical Research Center, Silver Spring, Maryland, United States
- Noguchi Memorial Institute of Medical Research, Legon, Ghana